CLINICAL TRIAL: NCT06867809
Title: Pilot Study to Evaluate the Safety and Tolerability of Spinal Cord Stimulation (SCS) and Paired Spine And Brain Stimulation For Movement Recovery After Spinal Cord Injury (SCI)
Brief Title: Spine and Brain Stimulation for Movement Recovery After Cervical Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jason Carmel (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Jason Carmel, Associate Professor of Neurology, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV3409; 5UE5NS070697-15 (NIH)
Record Dates: First submitted 2025-02-27; First posted 2025-03-10 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Spinal Cord Injury; Spinal Cord Injury Cervical
Keywords: Spinal Cord Injury; Spinal Cord Stimulation; Neurorehabilitation; Neurological Recovery
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Masking Description: Given that this is a single-arm, open label study, complete masking is not possible. However, to the greatest extent possible, subjects will be blinded to the stimulation-on versus stimulation-off conditions during assessments. In support of the blind, the stimulation condition will be determined by randomization, and both the subjects and the assessors will be blinded to the assignment of the stimulation condition. The stimulation-on condition will begin with a gradual ramp up of stimulation over the course of a minute as subjects are known to acclimate to the presence of stimulation relatively quickly; likewise, the stimulation-off condition will begin with the same one-minute ramp up of stimulation followed by a ramp down of stimulation to off over one minute.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Epidural Spinal Cord Stimulation (Experimental): Participants will undergo temporary placement of cervical epidural spinal cord stimulation (SCS) electrodes. They will undergo 2 visits of stimulation optimization based on mapping of motor responses to SCS and clinical assessments at a range of SCS parameters. Once a stimulation plan has been established, subjects will undergo baseline assessments with and without SCS over 2 visits. Subjects will then undergo 15 days of continuous SCS in conjunction with structured rehabilitation with occupational therapy. On each day of therapeutic stimulation, subjects will receive two sessions of SCS plus structured rehabilitation (for up to 1.5 hours per session). Subjects will undergo a clinical assessment with and without stimulation at the midpoint of the therapeutic stimulation period. After this therapeutic stimulation period, subjects will undergo 2 days of repeat assessments.
  Interventions: Device: Epidural spinal cord stimulation and paired spine and brain stimulation

INTERVENTIONS:
Device: Epidural spinal cord stimulation and paired spine and brain stimulation — The spinal cord and brain stimulator allows for stimulation of the spinal cord and brain. Spinal cord stimulation (SCS) is provided by temporarily implanted SCS catheter electrode leads (Medtronic) that are connected to an external stimulator (Digitimer); brain stimulation is provided by transcranial magnetic stimulation (TMS).

SUMMARY:
Stimulation of the spinal cord and brain represents a new experimental therapy that may have potential to restore movement after spinal cord injury. While some scientists have begun to study the effect of electrical stimulation on patient's ability to walk and move their legs after lower spinal cord injury, the use of stimulation of the upper (cervical) spine to restore arm and hand function after cervical spinal cord injury remains less well explored. The investigators are doing this research study to improve understanding of whether cervical spinal cord stimulation and brain stimulation can be used to improve arm and hand function. To do this, the investigators will combine spine stimulation (in the form of electrical stimulation from electrical stimulation wires temporarily implanted next to the cervical spinal cord) and brain stimulation (in the form of transcranial magnetic stimulation). The investigators will perform a series of experiments over 29 days to study whether these forms of stimulation can be applied and combined to provide improvement in arm and hand function.

DETAILED DESCRIPTION:
Loss of movement following spinal cord injury (SCI) often results from incomplete disruption of structures within the spinal cord, leaving some residual pathways of communication intact. Epidural spinal cord stimulation (SCS) has been used to recruit these residual communication pathways' spared circuits and restore walking in patients with leg paralysis. But SCS to improve arm and hand function remains largely unexplored, even though this is the commonest type of SCI and restoration of upper limb function is of highest priority to patients. The goal of this study is to understand the interactions between SCS and residual neural communication pathways in the brain and spine that control arm and hand function in order to restore movement after cervical SCI.

This is a pilot study in which patients with traumatic spinal cord injury will undergo temporary placement of small electronic stimulation wires near the cervical spinal cord followed by a series of experiments over 29 days focused on three main aims. In Aim 1 (mapping responses to SCS), the investigators will map patient's motor responses to SCS to identify how motor responses are affected by areas of spinal cord injury. In Aim 2 (pairing SCS with attempted motor activation and brain stimulation), the investigators will combine SCS with patient attempts to move in order to study how SCS interacts with conscious motor control and also pair SCS with brain stimulation using transcranial magnetic stimulation. Finally, in Aim 3 (therapeutic effects), the investigators seek to use SCS to change the natural electrical circuits in the spinal cord and observe changes in motor function in both the short- and long-term.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years with incomplete traumatic SCI (American Spinal Injury Association (ASIA) B-D, levels between C4 to T1) incurred > 1 year before the start of the study
* At least 2/5 motor power in at least one upper extremity muscle group
* International Standards for Neurological Classification of Spinal Cord Injury Upper Extremity Motor Score (ISNCSCI-UEMS) ≤ 40/50
* Able to follow multistep commands
* Ability and willingness to provide informed consent
* English speaking

Exclusion Criteria:

* Cervical or thoracic stenosis that would preclude safe lead placement
* Any ongoing ventilator use (continuous or intermittent)
* Urinary tract infection or pneumonia requiring treatment (within past 3 months)
* Skin ulcers or other lesions
* History of posterior cervical fusion
* Autonomic dysreflexia requiring treatment (within past 3 months)
* Implanted brain stimulators
* Intracranial aneurysm clips
* Ferromagnetic metallic implants in the head (except for within mouth)
* Any active implanted device including intrathecal medication pumps or existing spinal cord stimulators (does not include non-active spinal instrumentation such as rods, screws, or interbody devices)
* Cochlear implants
* Cardiac pacemaker/defibrillator
* Any history of seizures
* Family history of idiopathic epilepsy in a first degree relative
* Bipolar disorder
* Any history of suicide attempt
* Active psychosis
* Intracranial lesion or increased intracranial pressure
* History of stroke or intracranial neurologic conditions with structural damage
* Medications that lower seizure threshold
* Substance use that lowers seizure threshold (heavy alcohol use)
* Moderate to severe heart disease
* Pregnancy or plans to become pregnant within the study period
* Any other medical or psychological condition that precludes involvement in the study as determined by a study physician

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Serious adverse events related to the study device | From enrollment to the end of follow up at 30 weeks
  To assess safety of spinal cord stimulation and paired spine and brain stimulation for movement recovery after spinal cord injury, the investigators will record the number of serious adverse events related to the study device.
Cessation of spinal cord stimulation or brain stimulation due to participant request | From enrollment to the end of follow up at 30 weeks
  To assess tolerability of spinal cord and brain stimulation for movement recovery after spinal cord injury, the investigators will record the number of instances a participant requests permanent cessation of stimulation.

SECONDARY OUTCOMES:
Efficacy derived from spine-only and brain-only recruitment curves | Compared at visit 7/8 to visit 24/25 (~end of week 2 and end of week 5)
  Efficacy of stimulation is calculated as 1/threshold for provoking an motor evoked potentials. The threshold will be calculated from the spine-only and brain-recruitment curves. It is measured in units of 1/mA.
Selectivity derived from spine-only and brain-only recruitment curves | Compared at visit 7/8 to visit 24/25 (~end of week 2 and end of week 5)
  Selectivity of stimulation is calculated from the recruitment curves of the target muscle compared to non-targeted muscles. Selectivity is unitless.
Immediate effect of volitional motor activation combined with spinal stimulation | Compared at visit 7/8 to visit 24/25 (~end of week 2 and end of week 5)
  Immediate effect of volitional motor activation combined with spinal stimulation will be defined as the area under the curve (AUC) of the motor evoked potential (MEP) generated by attempted volitional activation optimally integrated with SCS divided by the sum of MEPs generated by attempted volitional activation at 10%-20% maximum effort alone and SCS alone. The immediate effect is unitless.
Immediate pairing effect of spine and brain stimulation | Compared at visit 7/8 to visit 24/25 (~end of week 2 and end of week 5)
  Immediate pairing effect of spine and brain stimulation will be defined as the area under the curve (AUC) of the motor evoked potential (MEP) generated by optimally paired spine and brain stimulation divided by the sum of MEPs generated by SCS and TMS alone. Immediate pairing effect is unitless.
Lasting effects of sustained spine and brain pairing | Compared at visit 7/8 to visit 24/25 (~end of week 2 and end of week 5)
  To analyze the effects of sustained pairing (facilitation of muscle responses to spine and/or brain stimulation following sustained pairing), the AUC of target muscle MEPs generated from spine-only and brain-only stimulation will be compared before sustained pairing, immediately after, and every 15 minutes for up to an hour. AUC of the MEP is measured in microVolt-seconds.
Magnitude of motor evoked potentials in TMS maps | Compared at visit 7/8 to visit 24/25 (~end of week 2 and end of week 5)
  Magnitude of motor evoked potentials (MEPs) are calculated as the area under the curve of the MEP. The unit of the AUC of the MEP is microVolt-seconds. These values are then weighted across the area of responsive cortex. The final unit of measure is microVolt-seconds-cm^2.
Size of responsive cortex in TMS maps | Compared at visit 7/8 to visit 24/25 (~end of week 2 and end of week 5)
  The size of the responsive cortex will be measured as an area of responsive cortex. The unit of measure is cm^2.
Power of cortical field potentials from EEG | Compared with and without stimulation at visit 7/8 to visit 24/25 (~end of week 2 and end of week 5)
  Power of cortical field potentials will be calculated from EEG using the Hilbert transform. The units of power are micro-Volts-squared per Hz.
Canadian Occupational Performance Measure (COPM)- Task Importance | Compared with and without stimulation at visits 7/8, 16, and 24/25 (~end of week 2, beginning of week 4, and end of week 5)
  The COPM is a standard subjective assessment in occupational therapy. In this assessment, participants identify a list of daily tasks (including in areas of self-care, leisure, etc) that are important to them, rank the importance of that task to them (1-10, 10 being most important).
Canadian Occupational Performance Measure (COPM)- Self-perception of performance | Compared with and without stimulation at visits 7/8, 16, and 24/25 (~end of week 2, beginning of week 4, and end of week 5)
  The COPM is a standard subjective assessment in occupational therapy. In this assessment, participants identify a list of daily tasks (including in areas of self-care, leisure, etc) that are important to them, rank their self-perception of their performance of that task (1-10, 10 being best performance).
Canadian Occupational Performance Measure (COPM)- Self-perception of satisfaction | Compared with and without stimulation at visits 7/8, 16, and 24/25 (~end of week 2, beginning of week 4, and end of week 5)
  The COPM is a standard subjective assessment in occupational therapy. In this assessment, participants identify a list of daily tasks (including in areas of self-care, leisure, etc) that are important to them, then rank their self-perception of their satisfaction with their performance of that task (1-10, 10 being highest satisfaction).
Patient Global Impression of Change | Study visit 25 (~end of week 5)
  The Patient Global Impression of Change provides a broad assessment of the patient or clinician's response to a therapy. Using a 7-point Likert scale ranging from (1) very much improved to (7) very much worse, patients are asked to rate their overall status with respect to their spinal cord injury since starting the therapy in the trial. The investigators will record the numerical value of the participant's answer to the 7-point Likert scale questionnaire.
Clinician Global Impression of Change | Study visit 25 (~end of week 5)
  The Clinician Global Impression of Change provides a broad assessment by the clinician of the patient's response to a therapy. Using a 7-point Likert scale ranging from (1) very much improved to (7) very much worse, clinicians are asked to rate the patient's overall status with respect to their spinal cord injury since starting the therapy in the trial. The investigators will record the numerical value of the participant's answer to the 7-point Likert scale questionnaire.
Off Target Effects Questionnaire | Study visit 25 (~end of week 5)
  The Off Target Effects Questionnaire asks the participant simple yes/no questions about the impact of cervical stimulation on a number of other functions outside of arm and hand function including spasticity, bowel/bladder function, sexual function, balance, and cognition). The questionnaire also invites the participant to describe any changes in each of these functions in free text form. Participants will record the yes/no and narrative answers to the questionnaire. The investigators will record and report the number of participants who complete the questionnaire.
Patient-specific Daily Activity Assessment | Compared with and without stimulation at visits 7/8, 16, and 24/25 (~end of week 2, beginning of week 4, and end of week 5)
  The Patient-specific Daily Activity Assessment is an outcome measure that will be developed individually for each participant based on their specific goals for recovery. Despite the variability across participants in specific content of this outcome measure, each one will be a quantitative metric of patient performance (e.g. for a participant who wishes to improve their time required to transfer out of a wheelchair, this assessment may be "time required to transfer from wheelchair to chair"). Percentage change in this outcome measure will be reported for each participant for the sake of comparison across individuals.
Grasp force | Compared with and without stimulation at visits 7/8, 16, and 24/25 (~end of week 2, beginning of week 4, and end of week 5)
  Grasp force will be measured with a manual dynamometer and reported in Newtons.
Pinch force | Compared with and without stimulation at visits 7/8, 16, and 24/25 (~end of week 2, beginning of week 4, and end of week 5)
  Pinch force will be measured with a manual dynamometer and reported in Newtons.
Box and block test score | Compared with and without stimulation at visits 7/8, 16, and 24/25 (~end of week 2, beginning of week 4, and end of week 5)
  In the box and block assessment, a subject is provided with one hundred and fifty 2.5 cm-sided blocks and asked to move as many of them as possible from one compartment (i.e. box) to another within 60 seconds. The box and block test provides an assessment of reach, grasp, transport, and release as well as fine motor control, coordination, and dexterity. The investigators will report the number of blocks moved successfully from one compartment to the other in 60 seconds.
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) score- Motor | Compared with and without stimulation at visits 7/8 and 24/25 (~end of week 2 and end of week 5)
  International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Scale (ISNCSCI-UESS) includes an assessment of motor and sensory function used to assess the severity of spinal cord injury. Motor scores characterize motor power in the bilateral upper and lower extremities (10 myotomes on each side) using the Medical Research Council (MRC) scale from grade 0 (no contraction) to grade 5 (normal). The maximum ISNCSCI motor score is 100. For motor scores, a higher score indicates better function.
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) score- Sensory | Compared with and without stimulation at visits 7/8 and 24/25 (~end of week 2 and end of week 5)
  International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Scale (ISNCSCI-UESS) includes an assessment of motor and sensory function used to assess the severity of spinal cord injury. Sensory scores include an assessment of light touch and pinprick for each of 28 dermatome bilaterally. For both light touch and pinprick, each bilateral dermatome is scored as follows: 0 for absent sensation, 1 for altered, and 2 for normal. The maximum sensory score is 224. For sensory scores, a higher score indicates better function.
International Standards for Neurological Classification of Spinal Cord Injury-Upper Extremity Measurement Scale (ISNCSCI-UEMS) | Compared with and without stimulation at visits 7/8, 16, and 24/25 (~end of week 2, beginning of week 4, and end of week 5)
  The ISNCSCI-UEMS is a subscore of the broader ISNCSCI assessment. The ISNCSCI-UEMS characterizes motor power in the bilateral upper extremities (5 myotomes on each side) using the Medical Research Council (MRC) scale from grade 0 (no contraction) to grade 5 (normal). The maximum ISNCSCI-UEMS score is 50. A higher score indicates better motor function.
Threshold to detect passive motion (TTDPM) | Compared with and without stimulation at visit 6 (~end of week 2)
  Proprioceptive function with and without continuous stimulation will be assessed using the threshold to detect passive motion (TTDPM) assessment at the metacarpophalangeal joint of the index fingers and at the joint located in a dermatome that corresponds to the primary site of stimulation. This outcome measure will be reported as the angle of motion (degrees) required to detect passive motion.
Graded Redefined Assessment of Strength, Sensation and Prehension (GRASSP)- Strength | Compared with and without stimulation at visits 7/8 and 24/25 (~end of week 2 and end of week 5)
  The Graded Redefined Assessment of Strength, Sensation and Prehension (GRASSP) is a validated assessment of sensorimotor function in patients with cervical spinal cord injury. The GRASSP (version 2) will be administered by an occupational therapist certified in GRASSP assessment. The GRASSP is reported as a series of subscores: strength (0-100, with 100 representing normal function).
Graded Redefined Assessment of Strength, Sensation and Prehension (GRASSP)- Sensation | Compared with and without stimulation at visits 7/8 and 24/25 (~end of week 2 and end of week 5)
  The Graded Redefined Assessment of Strength, Sensation and Prehension (GRASSP) is a validated assessment of sensorimotor function in patients with cervical spinal cord injury. The GRASSP (version 2) will be administered by an occupational therapist certified in GRASSP assessment. The GRASSP is reported as a series of subscores: sensation (0-24, with 24 representing normal sensation).
Graded Redefined Assessment of Strength, Sensation and Prehension (GRASSP)- Prehension Ability | Compared with and without stimulation at visits 7/8 and 24/25 (~end of week 2 and end of week 5)
  The Graded Redefined Assessment of Strength, Sensation and Prehension (GRASSP) is a validated assessment of sensorimotor function in patients with cervical spinal cord injury. The GRASSP (version 2) will be administered by an occupational therapist certified in GRASSP assessment. The GRASSP is reported as a series of subscores: prehension ability (0-24, with 24 representing normal function).
Graded Redefined Assessment of Strength, Sensation and Prehension (GRASSP)- Prehension Performance | Compared with and without stimulation at visits 7/8 and 24/25 (~end of week 2 and end of week 5)
  The Graded Redefined Assessment of Strength, Sensation and Prehension (GRASSP) is a validated assessment of sensorimotor function in patients with cervical spinal cord injury. The GRASSP (version 2) will be administered by an occupational therapist certified in GRASSP assessment. The GRASSP is reported as a series of subscores: prehension performance (0-40, with 40 representing normal prehension performance).
Capabilities of Upper Extremity Test (CUE-T) | Compared with and without stimulation at visits 7/8 and 24/25 (~end of week 2 and end of week 5)
  The Capabilities of Upper Extremity Test (CUE-T) is a validated assessment of sensorimotor function in patients with cervical spinal cord injury. The CUE-T will be administered by an occupational therapist certified in CUE-T assessment. The maximum CUE-T score is 124, with a higher score representing greater upper extremity function and a lower score representing greater limitations in upper extremity function.
Portion of study visits completed | From enrollment to the end of follow up at 30 weeks
  The investigators will record the portion of study visits completed and report this value as a percentage of total planned visits.

CONTACTS AND LOCATIONS:
Overall Officials: Jason B. Carmel, MD, PhD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - NewYork-Presbyterian Hospital / Columbia University Irving Medical Center (NYPH/CUIMC), New York, New York
  - NewYork-Presbyterian Allen Hospital / Columbia University Irving Medical Center (NYPH/CUIMC), New York, New York

IPD SHARING:
Plan to Share IPD: No